CLINICAL TRIAL: NCT07227090
Title: Mental Health Matters After Trauma Injury Survey
Brief Title: 2025 Mental Health Education Tool
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Bernard (Other)
Responsible Party: Sponsor-Investigator, Andrew Bernard, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 107433
Record Dates: First submitted 2025-11-05; First posted 2025-11-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Injury Traumatic; Mental Health Issue
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Survey patients who will not receive the mental health education document
- Health Education Document (Experimental): Survey patients who have been given the mental health education document
  Interventions: Behavioral: Mental Health Education Tool

INTERVENTIONS:
Behavioral: Mental Health Education Tool — A one-page mental health educational document provided to patients that have experienced trauma injury. The document provides brief evidence-based mindfulness practices in stress reduction, as well as information on how and when to address mental health issues.
  Arms: Health Education Document

SUMMARY:
The goal of this study is to learn if implementing a mental health educational resource handout will affect patient confidence, awareness, and knowledge of how to address mental health after trauma injury.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adult trauma patients

Exclusion Criteria:

* Participant less than 18 years old
* Non-English speaking or need of translator
* Subject doesn't complete survey

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Participant confidence in accessing mental health resources | Baseline
  Survey question with Likert type scale from 1 - 10 with higher scores indicating greater confidence
Participant confidence in receiving mental health support | Baseline
  Survey question with Likert type scale from 1 - 10 with higher scores indicating greater confidence

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bernard, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No